CLINICAL TRIAL: NCT02997566
Title: Autonomic Modulation and Facial Expression in Autism Spectrum Disorder: Cross-sectional Study
Brief Title: Autonomic Modulation and Facial Expression in Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luiz Carlos Marques Vanderlei, PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Other Study IDs: 57347916.5.0000.5402
Record Dates: First submitted 2016-12-15; First posted 2016-12-20 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Autistic Disorder; Autism Spectrum Disorder
Keywords: Autonomic Nervous System; Sympathetic Nervous System; Heart Rate
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Autistic Disorder: Age: 3 to 14 years-old Gender: male and female Autism Spectrum Disorder
  Interventions: Other: Autonomic evaluation
- Typical: Age: 3 to 14 years-old Gender: male and female Typical
  Interventions: Other: Autonomic evaluation

INTERVENTIONS:
Other: Autonomic evaluation

SUMMARY:
Background: the autism spectrum disorders (ASD) can be related with abnormalities in cortical structures and cause behavior imbalances. In addition, as soon as the diagnosis is done, the better will be the prognosis. In this context, heart rate variability (HRV) stands out, which is a non-invasive tool representing autonomic modulation, with potential prognostic value. The literature showed there are no changes in HRV at rest using linear methods of analysis, but changes can be identified during tasks. Nonlinear methods of HRV are more sensitive and provide additional information to the linear. Objective: to analyze autonomic modulation using nonlinear and linear indexes of HRV in children with ASD at rest and during tasks in comparison to typical children. In addition, to correlate HRV analysis between them, also between behavior and severity of the disease. Methods: this study involves both typical children and children with ASD. Autonomic modulation will be performed using nonlinear indices (extracted from Poincaré plot, detrended fluctuation of tendency analysis and recurrence plot) and linear indices of HRV in the time (RMSSD e SDNN) and frequency domain (LF, HF, VLF). The tasks consist in games to identify and recognize faces and facial expressions. Behavior and severity of the disease will be evaluated using the Autism Behavior Checklist and the Childhood Autism Rating Scale respectively. Statistical Analysis: to identify differences between moments and protocols two-way analysis of variance will be used along with the Bonferroni post-test or Dunn post-test according to the data distribution. Statistical significance will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Children with autistic disorder or typical development.

Exclusion Criteria:

* Participants that do not participant of all evaluations.
* Participants with an error superior to 5% in the RR intervals series.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with autistic disorder or typical development.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Autonomic evaluation | June, 2017
  Heart rate variability at rest, during facial expression games and finish at rest.

SECONDARY OUTCOMES:
Childhood Autism Rating Scale (CARS) | June, 2017
Autistic Behavior Checklist | June, 2017

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos M Vanderlei, PhD, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Universidade Estadual Paulista Júlio de Mesquita Filho, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided